CLINICAL TRIAL: NCT05232916
Title: A Randomized, Multicenter, Placebo-controlled, Phase 3 Study to Evaluate the Efficacy and Safety of HER2/Neu Peptide GLSI-100 (GP2 + GM-CSF) in HER2/Neu Positive Subjects With Residual Disease or High-Risk PCR After Both Neoadjuvant and Postoperative Adjuvant Trastuzumab-based Therapy (FLAMINGO-01)
Brief Title: Phase 3 Study to Evaluate the Efficacy and Safety of HER2/Neu Peptide GLSI-100 (GP2 + GM-CSF) in HER2/Neu Positive Subjects
Acronym: FLAMINGO-01
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Greenwich LifeSciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLSI-21-01
Record Dates: First submitted 2022-01-31; First posted 2022-02-10 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: HER2/neu positive; Residual disease; pCR; Extended adjuvant; GP2; Immunotherapy; HLA type
MeSH Terms: conditions — Breast Neoplasms; Neoplasm, Residual

STUDY DESIGN:
Intervention Model Description: HLA-A*02 subjects will be randomized to GLSI-100 or placebo. Treatment consists of 6 intradermal injections, Primary Immunization Series (PIS), over the first 6 months of treatment and 5 booster intradermal injections spaced 6 months apart. A third open-label arm will explore GLSI-100 immunotherapy in non-HLA-A*02 positive and HER2/neu positive subjects.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- 0.9% Normal Saline (Placebo Comparator): 0.9% normal saline in HLA-A*02 positive and HER2/neu positive subjects administered intradermally every month for first 6 months then every 6 months for next 2.5 years (11 intradermal injections over 3 years)
  Interventions: Biological: Placebo
- GLSI-100 (Experimental): GLSI-100 immunotherapy in HLA-A*02 positive and HER2/neu positive subjects administered intradermally every month for first 6 months then every 6 months for next 2.5 years (11 intradermal injections over 3 years)
  Interventions: Biological: GLSI-100
- GLSI-100, Open-label (Experimental): Open-label arm: GLSI-100 immunotherapy in non-HLA-A*02 positive and HER2/neu positive subjects administered intradermally every month for first 6 months then every 6 months for next 2.5 years (11 intradermal injections over 3 years)
  Interventions: Biological: GLSI-100

INTERVENTIONS:
Biological: Placebo — 0.9% Normal Saline
  Arms: 0.9% Normal Saline
Biological: GLSI-100 — 500 mcg/mL GP2 and 125 mcg/mL GM-CSF
  Arms: GLSI-100; GLSI-100, Open-label

SUMMARY:
This is a prospective, randomized, double-blinded, placebo-controlled, multi-center, Phase 3 study of GLSI-100 immunotherapy in HLA-A*02 positive and HER2/neu positive subjects who are at high risk for disease recurrence and have completed both neoadjuvant and postoperative adjuvant standard of care therapy. Treatment consists of 6 intradermal injections, Primary Immunization Series (PIS), over the first 6 months of treatment and 5 booster intradermal injections spaced 6 months apart. A third open-label arm will explore GLSI-100 immunotherapy in non-HLA-A*02 positive and HER2/neu positive subjects.

ELIGIBILITY:
Inclusion Criteria:

* HLA-A*02-positive, unless being enrolled in the third non-HLA-A*02 arm
* Histologically confirmed diagnosis of HER2/neu positive primary breast cancer for all tumors biopsied (multifocal, multicentric, or synchronous contralateral disease)
* Completion of both neoadjuvant and adjuvant trastuzumab-based standard of care breast cancer therapy
* Stage I, II, or III at presentation with pathologic evidence of residual invasive carcinoma in the breast or axillary lymph nodes (residual disease) at surgery following completion of neoadjuvant therapy -OR- Stage III at presentation with pathologic complete response (pCR) at surgery following completion of neoadjuvant therapy
* The subject can begin study therapy within one year of completion of adjuvant trastuzumab-based therapy and any other standard therapies, but, study therapy can be administered concurrently with endocrine therapy.
* No clinical evidence of residual or persistent breast cancer per treating physician assessment
* ECOG 0-2
* Adequate organ function
* Negative pregnancy test or evidence of post-menopausal status
* If of childbearing potential, willing to use a form of highly effective contraception
* Subject must both reside in and have been treated for their cancer in the country in which the clinical site is located.

Exclusion Criteria:

* Stage IV cancer or metastatic breast cancer at any time
* Inflammatory breast cancer
* Receiving other investigational agents
* Receiving chemotherapy
* Requiring long-term systemic treatment with corticosteroids or other immunosuppressive therapy
* History of immunodeficiency or active autoimmune disease
* A history of serious allergic reactions, including anaphylaxis, to human granulocyte-macrophage colony-stimulating factors such as sargramostim, yeast-derived products, or any component of the investigational product
* Other malignancies except adequately treated in situ carcinoma of the cervix or basal cell or squamous cell carcinoma of the skin
* Active infection
* Known HIV infection with a detectable viral load within 6 months of the anticipated start of treatment. Note: Subjects on effective antiretroviral therapy with an undetectable viral load within 6 months of the anticipated start of treatment are eligible for this trial.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2022-08-11 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Invasive Breast Cancer-free Survival (IBCFS) | Median 4 years of follow-up (interim analysis planned)
  IBCFS is defined as the time from the first dose of study medication until the date of ipsilateral invasive breast cancer recurrence, ipsilateral local-regional invasive breast cancer recurrence, distant recurrence, contralateral invasive breast cancer, or any cause mortality.

SECONDARY OUTCOMES:
Invasive Disease-free Survival (IDFS) | Median 4 years of follow-up (interim analysis planned)
  IDFS is defined as the time from the first dose of study medication until the date of ipsilateral invasive breast cancer recurrence, ipsilateral local-regional invasive breast cancer recurrence, distant recurrence, contralateral invasive breast cancer, second primary non-breast invasive cancer, or any cause mortality.
Distant Disease-free Survival (DDFS) | Median 4 years of follow-up (interim analysis planned)
  DDFS will be defined as the time from the first dose of study medication to the time of distant disease recurrence or death.
Overall Survival | Median 4 years of follow-up (interim analysis planned)
  Overall survival will be defined as the time from the first dose of study medication until death from any cause.
Quality of Life Questionnaire Core 30 (QLQ-C30) | Baseline and 36 months
  European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire Core 30 (QLQ-C30)
Quality of Life FACT-GP5 | Baseline and 36 months
  FACT-GP5 to assess global side effect impact

OTHER OUTCOMES:
Immune Response Measurements | Screening, Baseline, Month 4, Month 6, Month 12, Month 13, Month 18, Month 24, Month 25, Month 30, Month 36, Month 37, Month 42, Month 48
  Immune response will be measured by Delayed-Type Hypersensitivity (DTH) tests and immunologic assays.

CONTACTS AND LOCATIONS:
Overall Officials: Mothaffar F Rimawi, MD, Principal Investigator — Baylor College of Medicine
Locations (161):
- United States (40):
  - Tucson Medical Center HealthCare - Tucson-Rudasill, Tucson, Arizona
  - Providence St. Jude Medical Center - Virginia K. Crosson Cancer Center, Fullerton, California
  - University of California San Diego - Moores Cancer Center, La Jolla, California
  - University of Southern California - Norris Comprehensive Cancer Center, Los Angeles, California
  - Stanford Medicine Cancer Center - Stanford Women's Cancer Center, Palo Alto, California
  - University of California San Francisco - Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of California Los Angeles - Hematology / Oncology Parkside, Santa Monica, California
  - PIH Health Hospital - Whittier Hospital, Whittier, California
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Yale Cancer Center - Smilow Cancer Hospital, New Haven, Connecticut
  - Johns Hopkins Medicine - Kimmel Cancer Center-Sibley Memorial Hospital, Washington D.C., District of Columbia
  - University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University - Northwestern Memorial Hospital, Chicago, Illinois
  - Maryland Oncology Hematology, Annapolis, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Minnesota Oncology, Maple Grove, Minnesota
  - Siteman Cancer Center - Washington University Medical Campus, St Louis, Missouri
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Nebraska Medicine - University of Nebraska Medical Center, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - Cooper University Health Care, Camden, New Jersey
  - New York Oncology Hematology, Albany, New York
  - New York-Presbyterian - Columbia University Irving Medical Center, New York, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - Oncology Hematology Care, Cincinnati, Ohio
  - Compass Oncology - Northwest Cancer Specialists, Tigard, Oregon
  - Redeemer Health - Holy Redeemer Hospital, Meadowbrook, Pennsylvania
  - Sidney Kimmel Comprehensive Cancer Center - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Texas Oncology - Austin, Austin, Texas
  - Texas Oncology - Dallas Presbyterian Hospital, Dallas, Texas
  - Texas Oncology - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine - Dan L. Duncan Comprehensive Cancer Center, Houston, Texas
  - The University of Texas Health Sciences Center at San Antonio - Mays Cancer Center, San Antonio, Texas
  - Texas Oncology - San Antonio, San Antonio, Texas
  - Texas Oncology - Gulf Coast, Sugar Land, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - University of Utah - Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Cancer Specialists, Fairfax, Virginia
- France (20):
  - Sainte-Catherine - Institut du Cancer Avignon-Provence (ICAP), Avignon
  - Clinique Pasteur-Lanroze, Brest
  - Centre François Baclesse (CLCC), Caen
  - Pôle Santé Léonard De Vinci, Chambray-lès-Tours
  - Centre Hospitalier de Cholet, Cholet
  - Centre Hospitalier Alpes Leman, Contamine-sur-Arve
  - Centre Léon Bérard, Lyon
  - Hôpital Privé du Confluent, Nantes
  - Centre Hospitalier Privé Sainte-Marie Osny, Osny
  - Institut Curie, Paris
  - Hospices Civils de Lyon, Pierre-Bénite
  - Hôpital NOVO (Nord-Ouest Val-d'Oise), Pontoise
  - Institut Jean Godinot (CLCC), Reims
  - Institut Curie, Saint-Cloud
  - Centre Hospitalier Privé Saint-Grégoire, Saint-Grégoire
  - Centre Hospitalier Universitaire de Saint-Étienne, Saint-Priest-en-Jarez
  - Institut de cancérologie Strasbourg Europe, Strasbourg
  - Hôpital Privé Drôme Ardèche, Valence
  - Hôpital Robert Schuman, Vantoux
  - Institut Gustave Roussy, Villejuif
- Germany (38):
  - Haematologie-Onkologie im Zentrum MVZ GmbH, Augsburg
  - Klinikum Bayreuth GmbH, Bayreuth
  - DBZ Onkologie GmbH, Berlin
  - Helios Klinikum Berlin-Buch GmbH, Berlin
  - Marienhospital Bottrop gGmbH, Bottrop
  - Evangelisches Diakonie-Krankenhaus gGmbH, Bremen
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Städtisches Klinikum Dessau, Dessau
  - St.-Johannes Hospital Dortmund, Dortmund
  - Universitaetsklinikum Carl Gustav Carus Dresden an der Technischen Universitaet Dresden AöR, Dresden
  - MVZ Medical Center Duesseldorf GmbH, Düsseldorf
  - Studienzentrale für das MVZ Eggenfelden e.K., Eggenfelden
  - Evangelisches Kliniken Essen-Mitte gGmbH, Essen
  - Klinikum Frankfurt Höchst GmbH, Frankfurt
  - Praxis für Interdisziplinäre Onkologie und Haematologie GbR, Freiburg im Breisgau
  - Helios Klinikum Gifhorn GmbH, Gifhorn
  - Universitätsmedizin Göttingen, Göttingen
  - Krankenhaus St. Elisabeth und St. Barbara Halle (Saale) GmbH, Halle
  - Mammazentrum Hamburg MVZ GbR, Hamburg
  - Gynäkologische Praxisklinik Hamburg-Harburg, Harburg
  - National Center For Tumor Diseases (NCT) Heidelberg, Heidelberg
  - Elisabeth Krankenhaus GmbH, Kassel
  - MVZ GynKrefeld GmbH, Krefeld
  - Gemeinschaftspraxis für Hämatologie und Onkologie Langen, Langen
  - Studienzentrum UnterEms Leer, Leer
  - RKH Klinken Ludwigsburg-Bietigheim gGmbH, Ludwigsburg
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz KöR, Mainz
  - Heidelberg University, Mannheim
  - Klinikum der Technischen Universitaet Muenchen (TUM Klinikum), Munich
  - München Klinik gGmbH, Munich
  - Klinikum Südstadt Rostock Eigenbetrieb der Hanse und Universitätsstadt Rostock, Rostock
  - Gesundheits und Pflegezentrum Ruesselsheim gGmbH, Rüsselsheim am Main
  - Diakonissen-Stiftungs-Krankenhaus Speyer, Speyer
  - Klinikum Mutterhaus der Borromäerinnen gGmbH, Trier
  - Universitätsklinikum Ulm AöR, Ulm
  - Marienhospital Witten, Witten
  - Klinikum Worms gGmbH, Worms
  - Helios Universitätsklinikum Wuppertal, Wuppertal
- St. Vincent's University Hospital, Dublin, Ireland
- Italy (10):
  - Azienda Ospedaliero Universitaria di Bologna Policlinico di Sant'Orsola IRCCS (Istituto Di Ricerca E Di Cura A Carattere Scientifico), Bologna
  - Ospedale Policlinico San Martino IRCCS (Istituto Di Ricerca E Di Cura A Carattere Scientifico), Genova
  - Humanitas Research Hospital, Milan
  - Azienda Ospedaliera Universitaria Federico II Di Napoli, Naples
  - Istituto Nazionale Tumori Fondazione Pascale IRCCS (Istituto Di Ricerca E Di Cura A Carattere Scientifico), Naples
  - Azienda Ospedaliero Universitaria Maggiore della Carità di Novara, Novara
  - Istituto Oncologico Veneto, Padua
  - Istituti Clinici Scientifici Maugeri Spa Società Benefit IRCCS (Istituto Di Ricerca E Di Cura A Carattere Scientifico), Pavia
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Istituto Di Ricerca E Di Cura A Carattere Scientifico), Rome
- Poland (9):
  - Przychodnia Lekarska KOMED Roman Karaszewski, Konin
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej (ZOZ) Szpital Uniwersytecki w Krakowie, Krakow
  - Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie, Krakow
  - Samodzielny Publiczny Zakład Opieki Zdrowotnej (SPOZOZ) Opolskie Centrum Onkologii im. prof. Tadeusza Koszarowskiego w Opolu, Opole
  - Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan
  - Centrum Medyczne MrukMed, Rzeszów
  - Wojewodzki Szpital Specjalistyczny im. Janusza Korczaka w Słupsku, Słupsk
  - Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie, Warsaw
  - Wojskowy Instytut Medyczny, Państwowy Instytut Badawczy, Warsaw
- Romania (4):
  - Filantropia Clinical Hospital, Bucharest
  - Neolife Baneasa Bucharest Medical Center, Bucharest
  - Institute of Oncology "Prof Dr Ion Chiricuta", Cluj-Napoca
  - Oncomed SRL - Oncology Center, Timișoara
- Spain (39):
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Hospital General Universitario Dr. Balmis, Alicante
  - Hospital Universitario de Badajoz, Badajoz
  - Hospital Clínic De Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital San Pedro de Alcántara, Cáceres
  - Hospital Universitario Reina Sofía, Córdoba
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar
  - Hospital Universitario de Fuenlabrada, Fuenlabrada
  - Hospital Galdakao-Usansolo, Galdakao
  - Hospital Universitario Clínico San Cecilio, Granada
  - Hospital Universitario de Jaén, Jaén
  - Hospital Universitario de Jerez de la Frontera, Jerez de la Frontera
  - Hospital Universitari Arnau de Vilanova (Lleida), Lleida
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda
  - Althaia, Xarxa Assistencial Universitària de Manresa, Manresa
  - Hospital Clínico Universitario Virgen de la Victoria, Málaga
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna
  - Hospital Universitario Donostia, San Sebastián
  - Hospital Universitari General de Catalunya - Grupo Quirónsalud, Sant Cugat del Vallès
  - Hospital Universitario San Juan de Alicante, Sant Joan d'Alacant
  - Hospital Universitario Nuestra Señora de Candelaria, Santa Cruz de Tenerife
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario de Toledo, Toledo
  - Consorcio Hospital General Universitario de Valencia, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitari Arnau de Vilanova (Valencia), Valencia
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: No